CLINICAL TRIAL: NCT04119154
Title: Feasibility and Accuracy of Nanosensor-based Cancer Diagnosis at the Point-of-care (Chedza)
Acronym: Chedza
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Botswana Harvard AIDS Institute Partnership (Other); Massachusetts General Hospital (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Scott Dryden-Peterson, Research Associate, Harvard School of Public Health (HSPH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BHP0111; UH3CA202637 (NIH)
Record Dates: First submitted 2019-10-04; First posted 2019-10-08 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Breast Neoplasms; Lymphoma
MeSH Terms: conditions — Breast Neoplasms; Lymphoma

STUDY DESIGN:
Intervention Model Description: Cancer suspects will undergo standard diagnostic evaluation and novel diagnostic. Single arm.
Masking Description: No masking, open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard diagnosis and CEM platform (Experimental): Participants will receive standard diagnostic approach and assessment by CEM platform
  Interventions: Diagnostic Test: Contrast Microhalography (CEM)

INTERVENTIONS:
Diagnostic Test: Contrast Microhalography (CEM) — Fine needle aspirates evaluated by CEM device

SUMMARY:
Prospective feasibility and validation study of a novel, near-to-care modality for diagnosis of malignancy among cancer suspects.

DETAILED DESCRIPTION:
Prospective feasibility and validation study of a novel contrast microhalography (CEM) device for diagnosis of malignancy in Botswana. Consenting patients identified by their providers as requiring a fine needle aspirate (FNA) or percutaneous biopsy for assessment for possible lymphoma or breast cancer will undergo standard diagnostic procedure. Concurrently these patients will have additional FNA fluid tested using the portable novel nanosensor-based device (CEM). Diagnosis made from standard anatomic pathology, flow cytometry, and/or cytology will be compared with the diagnosis made using the CEM platform. Assessment of the feasibility and acceptability of the CEM platform will be performed. Assessment of training requirements for CEM platform will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Botswana citizen
* Age 18 years or older
* Able and willing to provide informed consent
* Undergoing diagnostic procedure for palpable abnormality (biopsy, node/mass resection, or fine-needle aspirate) for diagnosis of possible lymphoid malignancy or breast cancer

Exclusion Criteria:

* Involuntary incarceration (prison, jail, etc.)
* Procedures involving internal organs or locations expected to have elevated risk of complication
* Increased risk for severe bleeding as defined as known hemophilia or other bleeding disorder, use of anticoagulants in past week (not including aspirin or other NSAIDS), advanced liver disease, or other condition determined by clinician to significantly increase bleeding risk of procedure
* Known pregnancy
* Critical illness as defined by current intensive care admission, hypotension (systolic BP<100mmHg), hypoxemia (O2 saturation <94% on room air), or other condition determined by clinician to significantly decrease physiologic tolerance of procedure
* Other condition felt by the clinician performing procedure to significantly increase risk of procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Accuracy for diagnosis of non-Hodgkin lymphoma | Day 1, at time of diagnosis
  Accuracy (proportion of true positive and true negative out of total number assessed) of CEM in comparison with standard diagnostic approach.
Accuracy for diagnosis of invasive breast cancer | Day 1, at time of diagnosis
  Accuracy (proportion of true positive and true negative out of total number assessed) of CEM in comparison with standard diagnostic approach.
Time to diagnosis | Day 1, at time of diagnosis
  Time from diagnostic procedure to knowledge of test result by the treating clinician
Proficiency in testing using CEM platform | Day 1, At completion of training
  Proportion of personnel of varying laboratory experience and training modalities with proficiency using CEM platform

SECONDARY OUTCOMES:
Accuracy for sub-type diagnosis (aggressive vs. indolent) of non-Hodgkin lymphoma | Day 1, at time of diagnosis
  Accuracy (proportion of true positive and true negative out of total number non-Hodgkin lymphoma) of CEM in comparison with standard diagnostic approach.
Accuracy for molecular subtype diagnosis of invasive breast cancer | Day 1, at time of diagnosis
  Accuracy (proportion of true positive and true negative out of total number of invasive breast cancers), compared with standard diagnostic approach, for the molecular subtype diagnosis of invasive breast cancer into estrogen-receptor positive, triple-negative, and other estrogen-receptor negative categories.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Weissleder, MD, PhD, Principal Investigator — Massachusetts General Hospital; Scott Dryden-Peterson, MD, MSc, Principal Investigator — Botswana Harvard AIDS Institute, Harvard TH Chan School of Public Health, Brigham and Women's Hospital
Locations (1):
- Botswana Harvard AIDS Institute, Gaborone, Botswana

IPD SHARING:
Plan to Share IPD: Yes
Completely anonymized data can be shared to investigators following successful receipt of IRB approval (Botswana and US committees).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Following completion of primary analysis.
Access Criteria: Sharing following required IRB approval (Botswana and US).

DOCUMENTS (1):
  • Informed Consent Form (2019-07-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT04119154/ICF_000.pdf